CLINICAL TRIAL: NCT02915939
Title: The Residential Care Transition Module
Acronym: RCTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Johns Hopkins University (Other); NYU Langone Health (Other); Benjamin Rose Institute (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1511S80406
Record Dates: First submitted 2016-09-19; First posted 2016-09-27 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Family caregiving; Institutionalization; Residential long-term care; Placement; Psychosocial support; Dementia; Caregivers; Nursing homes; Assisted Living Facilities; Long-Term Care; Intervention Study; Psychosocial Support Systems; Social Support; Coping; COVID-19
MeSH Terms: conditions — Alzheimer Disease; Dementia; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): The Residential Care Transition Module (RCTM) includes six in-person consultation sessions over a 4-month period conducted by a trained Transition Counselor (TC) with a primary family caregiver (self-identified as the person most responsible for providing on-going assistance to the care recipient in a residential long-term care setting such (RLTC) such as a nursing home or assisted living memory care unit.
  Interventions: Behavioral: The Residential Care Transition Module
- Usual Care Group (No Intervention): The usual care control group will adjust for the social engagement provided to the Residential Care Transition Module (RCTM )treatment condition. The Transition Counselor (TC) will provide quarterly contact calls and the research coordinator will send a bi-annual project newsletter to all participants. If caregivers in the control group initiate contact with the TC for care needs, the TC will provide information and referral support.

INTERVENTIONS:
Behavioral: The Residential Care Transition Module — Residential Care Transition Module sessions focus on the experiences of the caregiver, the care recipient, and (potentially) other family members immediately following residential long-term care (RLTC) admission. The sessions are designed to establish a therapeutic rapport with the caregiver and the family; provide a safe environment to explore stressors; examine family relational dynamics as they relate to the RLTC placement decision itself as well as the roles different family members play in the life of the caregiver and relative in RLTC; identify new modes of communication to facilitate more effective interactions with other family members and care staff; and identify effective ways to advocate for improved quality of care for and quality of life of their relatives in RLTC.
  Arms: Treatment Group

SUMMARY:
Emerging research on family caregiving and institutionalization has emphasized that families do not disengage from care responsibilities following a relative's admission to residential long-term care settings. The Residential Care Transition Module (RCTM) provides 6 formal sessions of consultation (one-to-one and family sessions) over a 4-month period to those family caregivers who have admitted a cognitively impaired relative to a residential long-term care setting (nursing home, assisted living memory care unit). The proposed mixed method, randomized controlled trial will determine whether and how the RCTM decreases family caregivers' emotional and psychological distress, placement-related strain, and increases relative's transitions back to the community. The RCTM will fill an important clinical and research gap by evaluating a psychosocial intervention designed for families following RLTC placement to determine whether and how this approach can help families better navigate the residential care transitions of relatives with Alzheimer's disease or a related dementia.

DETAILED DESCRIPTION:
Emerging research on family caregiving and institutionalization has found that families do not disengage from care responsibilities following relatives' admissions to residential long-term care settings. Families instead remain involved in a spectrum of care activities ranging from instrumental activities of daily living to emotional support. Perhaps for these reasons, a number of studies have noted that caregiving stress, depression, or other key outcomes remain stable or sometimes increase following residential long-term care (RLTC) entry for certain types of caregivers. A few interventions have attempted to increase family involvement after institutionalization, but no rigorous studies have demonstrated that these interventions are effective in helping families navigate transitions to RLTC environments.

The Residential Care Transition Module (RCTM) provides 6 formal sessions of consultation (one-to-one and family sessions) over a 4-month period to those family caregivers who have recently admitted a relative to a RLTC setting. In this randomized controlled trial, family members who have admitted a cognitively impaired relative to a RLTC setting will be randomly assigned to the RCTM [(n = 120)] or a usual care control condition [(n = 120)]. A mixed methods analysis will be used to pursue the following aims: Specific Aim 1: Assess whether the RCTM yields statistically significant reductions in family members' primary subjective stress and negative mental health outcomes; Specific Aim 2) Determine whether family members who receive the RCTM will indicate statistically significant decreases in secondary role strains over a 12-month period when compared to usual care controls; Specific Aim 3) Determine whether RCTM family members report statistically significant decreases in residential care stress when compared to family members in the usual care control group; and Specific Aim 4) Delineate the mechanism of action of RCTM under conditions of high and low success by "embedding" qualitative components (30 semi-structured interviews) at the conclusion of the 12-month evaluation.

The proposed project will fill an important clinical and research gap by evaluating a psychosocial intervention designed for families following RLTC placement that determines whether and how the RCTM can help families better navigate the residential care transitions of cognitively impaired relatives.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of relatives who have received a physician's diagnosis of Alzheimer's disease or a related dementia (ADRD)
* Family caregivers who consider themselves the most involved in visiting and providing assistance to a relative experiencing a long-stay admission to an assisted living, nursing home, memory care, or other residential long-term care setting. Those who share the primary caregiving role equally are also eligible.
* Family caregivers must be English speaking, 21 years of age or older
* Family caregivers on psychotropic medications, such as anti-depressants or anti-psychotics, will be eligible if they have remained on a stable dosage for the last 3 months

Exclusion Criteria:

* Family caregivers who are participating in any other type of service that provides one-to-one psychosocial consultation specifically for caregiving (support group participation is not a deterrent to enrollment, nor is general counseling not specific to caregiving)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in care-related strain | 12 months
  A 7-item measure of care-related strain that assesses the stress family caregivers perceive as a result of having a relative in residential care
Change in burden: Zarit Burden Interview | 12 months
  A 7-item version of the Zarit Burden Interview
Change in stress: Perceived Stress Scale | 12 months
  The Perceived Stress Scale

SECONDARY OUTCOMES:
Quantitative measure of resilience to negative psychosocial effects of COVID-19 | 0, 1 and 4 months post-pandemic onset
  Compare trajectories of caregiver stress and well-being across the treatment and control groups using quantitative (survey) data to determine whether the RCTM provides benefits in the context of COVID-19.
Qualitative measure of resilience to negative psychosocial effects of COVID-19 | 0, 1 and 4 months post-pandemic onset
  Compare trajectories of caregiver stress and well-being across the treatment and control groups using qualitative (experiences) data to determine whether the RCTM provides benefits in the context of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E. Gaugler, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, School of Nursing, 6-153 Weaver-Densford Hall, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data supporting our findings will be shared on the National Archive of Computerized Data on Aging (NACDA).
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Zmora R, Statz TL, Birkeland RW, McCarron HR, Finlay JM, Rosebush CE, Gaugler JE. Transitioning to Long-Term Care: Family Caregiver Experiences of Dementia, Communities, and Counseling. J Aging Health. 2021 Jan;33(1-2):133-146. doi: 10.1177/0898264320963588. Epub 2020 Sep 29. PMID 32990494
- [Background] Gaugler JE, Statz TL, Birkeland RW, Louwagie KW, Peterson CM, Zmora R, Emery A, McCarron HR, Hepburn K, Whitlatch CJ, Mittelman MS, Roth DL. The ResidentialCare Transition Module: a single-blinded randomized controlled evaluation of a telehealth support intervention for family caregivers of persons with dementia living in residential long-term care. BMC Geriatr. 2020 Apr 15;20(1):133. doi: 10.1186/s12877-020-01542-7. PMID 32293314
- [Background] Mitchell LL, Albers EA, Birkeland RW, Peterson CM, Stabler H, Horn B, Cha J, Drake A, Gaugler JE. Caring for a Relative With Dementia in Long-Term Care During COVID-19. J Am Med Dir Assoc. 2022 Mar;23(3):428-433.e1. doi: 10.1016/j.jamda.2021.11.026. Epub 2021 Dec 17. PMID 34929196
- [Background] Gaugler JE, Mitchell LL. Reimagining Family Involvement in Residential Long-Term Care. J Am Med Dir Assoc. 2022 Feb;23(2):235-240. doi: 10.1016/j.jamda.2021.12.022. Epub 2021 Dec 29. PMID 34973167
- [Derived] Urbanski DP, Birkeland RW, Albers EA, Roth DL, Baker ZG, Gustavson AM, Yam H, Gaugler JE. Process evaluation of the residential care transition module. BMC Health Serv Res. 2025 Oct 27;25(1):1412. doi: 10.1186/s12913-025-13547-2. PMID 41146257

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT02915939/Prot_SAP_000.pdf